CLINICAL TRIAL: NCT02256241
Title: The Role of RING Ubiquitin Ligases in Biologic and Oncologic Processes in Tissues of Mesenchymal Origin
Acronym: RING UB LIGASE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Technion, Israel Institute of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 0180-14-RMB
Record Dates: First submitted 2014-07-29; First posted 2014-10-03 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Group 1: Trauma Operation for Otherwise Healthy Patients; Group 2: Primary Tumors of Mesenchymal Origin

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples Without DNA — 1. Bone marrow will be collected from othewise healthy patients undergoing orthopedic surgery - arthroplasty for the treatment of degenerative joint disease or traumatised patients. The bone marrow will be collected from disposable tissue that is removed during the normal sequence of the surgery.
  2. Collection of connective tissue from patients with malignancies of musculoskeletal origin. The tissue that will be used is part of the resected tumor specimens. The tissue will be used for:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- The role of RING ubiquitin ligases in osteogenic progenitors: Bone marrow (BM) will be collected from healthy patients undergoing orthopedic surgery. BM will be collected from disposable tissue that is removed during the normal sequence of the surgery.
- The role of RING ubiquitin ligases in musculoskeletal cancer: Collection of connective tissue from patients with tumors of musculoskeletal origin - a part of the resected tumor specimens.

SUMMARY:
Stage 1:

Bone marrow will be collected from otherwise healthy patients undergoing orthopedic surgery - arthroplasty for the treatment of degenerative joint disease or traumatised patients. The bone marrow will be collected from disposable tissue that is removed during the normal sequence of the surgery. These cells will be used for:

Establishment of the role of RING ubiquitin ligases in osteogenic progenitors proliferation and differentiation in culture.

I. To determine the levels of RING ubiquitin ligases mRNA and protein in differentiating human mesenchymal precursor cells: To test the correlation between levels of RING ubiquitin ligases and degree of osteogenic differentiation, we will extract mesenchymal precursor cells from the collected tissue and test the mRNA protein level of RING ubiquitin ligases upon induction of differentiation. Specifically, we will compare the levels of RING ubiquitin ligases before and after the initiation of differentiational stimulus in time dependent manner by western blot and real time PCR analysis.

II. To test the impact of specific RING ubiquitin ligases on differentiation of human mesenchymal precursor cells: to test the impact of RING ubiquitin ligases on the differentiation of mesenchymal precursor cell from the collected tissue by testing the expression of classical differentiational bone markers by flow cytometry (fibronectin, CD105) and by Alkaline phosphatase (ALP) activity assay. For this aim we developed both a constitutive and Dox-regulated conditional overexpression and shRNA lenti-viral systems that enables efficient modulation of these RING ubiquitin ligases level.

III. Determine the role of RING ubiquitin ligases in proliferation and survival of human mesenchymal precursor cells: Via inhibition or overexpression of ligases in mesenchymal progenitor cells we will test the role of these ligases in proliferation and survival of mesenchymal precursors by using MTT assay, Propidion-Iodid (PI) and tunnel assays in flow cytometry analysis.

Stage 2:

Collection of connective tissue from patients with malignancies of musculoskeletal origin. The tissue that will be used is part of the resected tumor specimens. The tissue will be used for:

The establishment of the role/s of RING ligases in musculoskeletal cancers using cell culture and in vivo activation. Test if the expression of selected positive candidates from stage 1 correlates with cancer development and progression in human-derived samples Independently of our mechanistic experiment we aim to determine the relevance of these ligases to human musculoskeletal cancers. As the first step we will screen primary tumor biopsies at the protein level correlates with cancer grade and prognosis. Toward this aim we recently generated a highly specific several anti-monoclonal antibodies in our laboratory as well use comercial available antibodies .

DETAILED DESCRIPTION:
Stage 1:

Bone marrow will be collected from otherwise healthy patients undergoing orthopedic surgery - arthroplasty for the treatment of degenerative joint disease or traumatised patients. The bone marrow will be collected from disposable tissue that is removed during the normal sequence of the surgery. These cells will be used for:

Establishment of the role of RING ubiquitin ligases in osteogenic progenitors proliferation and differentiation in culture.

I. To determine the levels of RING ubiquitin ligases mRNA and protein in differentiating human mesenchymal precursor cells: To test the correlation between levels of RING ubiquitin ligases and degree of osteogenic differentiation, we will extract mesenchymal precursor cells from the collected tissue and test the mRNA protein level of RING ubiquitin ligases upon induction of differentiation. Specifically, we will compare the levels of RING ubiquitin ligases RING ubiquitin ligases before and after the initiation of differentiational stimulus in time dependent manner by western blot and real time PCR analysis.

II. To test the impact of RING ubiquitin ligases on differentiation of human mesenchymal precursor cells: to test the impact of RING ubiquitin ligases on the differentiation of mesenchymal precursor cell from the collected tissue by testing the expression of classical differentiational bone markers by flow cytometry (fibronectin, CD105) and by Alkaline phosphatase (ALP) activity assay. For this aim we developed both a constitutive and Dox-regulated conditional RING ubiquitin ligases overexpression and shRNA lenti-viral systems that enables efficient modulation of RING ubiquitin ligases level.

III. Determine the role of RING ubiquitin ligases in proliferation and survival of human mesenchymal precursor cells: We will test the role of their in proliferation and survival of mesenchymal precursors by using MTT assay, Propidion-Iodid (PI) and tunnel assays in flow cytometry analysis.

Stage 2:

Collection of connective tissue from patients with malignancies of musculoskeletal origin. The tissue that will be used is part of the resected tumor specimens. The tissue will be used for:

The establishment of the role/s of RING ubiquitin ligases in musculoskeletal cancers using cell culture and in vivo.

I. Test the role of our in proliferation and survival in musculoskeletal cancers: Using our lentiviral systems we will test the biological impact of inhibition and overexpression in musculoskeletal neoplastic cells.

II. Test whether inhibition or overexpression of these ligases impacts the biology of musculoskeletal cancers.We will check if inhibition of these ligases in malignant cells of musculoskeletal origin by lenti-viral infections induces differentiation. Infected cells will be analyzed for expression of differentiational markers in flow cytometry and immunohistochemistry.

III. Test if expression of RING ubiquitin ligases correlates with cancer development and progression in human-derived samples Independently of our mechanistic experiment we aim to determine the relevance of RING ubiquitin ligases to human musculoskeletal cancers.

Patients consent will be signed after properly informed at time of pre-surgical preparation visit. In cases when pre-surgical visit is not held consent will be signed prior to the day of surgery.

ELIGIBILITY:
Group 1:

* Inclusion Criteria:
* Healthy patients undergoing orthopedic surgery - arthroplasty for the treatment of degenerative joint disease or traumatised patients.
* Exclusion Criteria:
* Any malignancy in the past or active infection.

Group 2:

* Inclusion Criteria:
* patients with malignancies of musculoskeletal origin.
* Exclusion Criteria:
* Any malignancy of unknown origin or malignancy of multiple origins or active infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Healthy patients undergoing orthopedic surgery - arthroplasty for the treatment of degenerative joint disease or traumatised patients.
  2. Patients with malignancies of musculoskeletal origin.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2014-10; Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Protein and mRNA levels of RING ubiquitin ligases during osteogenesis | 5 years
  To determine the levels of RING ubiquitin ligases mRNA and protein in differentiating human mesenchymal precursor cells. We will extract mesenchymal precursor cells from the collected tissue and test the mRNA and protein levels of RING ubiquitin ligases upon induction of differentiation.
Protein and mRNA levels of RING ubiquitin ligases in musculoskeletal tumors and its correlation to staging and grading | Time Frame: * 5 years
  It is not clear if RING ubiquitin ligases protein levels are elevated in soft tissue-derived cancers (primary and metastatic tumors) and whether there is a correlation between RING ubiquitin ligases levels and staging and grading of soft tissue-derived cancers. For this reason, we will check whether RING ubiquitin ligases expression correlates with cancer development and progression in human-derived samples. We will determine the relevance of RING ubiquitin ligases to human musculoskeletal cancers. To do this we will screen primary tumor biopsies for RNA and protein levels of RING ubiquitin ligases .

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam MC, Haifa, Israel